CLINICAL TRIAL: NCT01888913
Title: Patient Perspectives and Simulated Clinical Interactions
Brief Title: Patient Perspectives and Doctor Visits
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130158; 13-HG-0158
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Body Weight
Keywords: Body Weight; Virtual Environment; Natural History
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Women: Adult Women aged 18-50

SUMMARY:
Background:

- We are studying people s psychological experiences and how these relate to the way people respond have when they see information communicated in different ways. We are testing multiple research questions in this research.

Objectives:

- To learn about how to design future research studies. Also to learn about how to best give people information about health topics.

Eligibility:

- Women with a Body Mass Index of 25 or higher.

Design:

* Before the study visit, participants will answer some questions online about themselves, their experiences, and their thoughts about their weight.
* During the study visit, participants will watch a short scene from a movie, and then answer questions about it.
* Participants will have a simulated doctor visit with a computerized, virtual reality doctor. They will answer more questions about themselves, their experiences, and their thoughts about their weight. Then they will answer questions with researchers.

DETAILED DESCRIPTION:
The primary goal of this research project is to continue building an evidence base on the benefits or pitfalls of introducing genomic information into weight-related primary care encounters. We are particularly interested in how this information will impact patients health-related attitudes, beliefs and behavior, and patient perceptions of stigmatization. Furthermore, this project aims to determine whether a patient s emotional state during a clinical interaction will moderate the consequences of genomic information provision.

Genetic and genomic information are expected to be integrated into personalized prevention and treatment regimens of the future. Such information may influence patient beliefs, attitudes, and behaviors related to weight and obesity. Previous research has shown that provision of genomic information can lead to positive effects, negative effects and often no effect with respect to patient motivation for health-promoting behaviors. The literature describing the influence of emotion on judgment and decision-making suggests that patients emotional state may, in part, account for this discrepancy. By better understanding the influence of emotional state on patients reactions to general, weight-related genomic information, we may be better able to shape clinical communications of the future to increase the likelihood that genomic information will lead to positive, health-promoting behavior. Indeed, there is a need for exploration of strategies through which providers can counsel patients about weight such that patients feel motivated by the counseling, and that it does not make them feel stigmatized.

The current protocol describes two studies; both are randomized, controlled experiments. The first will be conducted through an internet panel via the Time-Sharing Experiments in the Social Sciences program. The current proposal was already reviewed and was successfully approved and funded for fielding through this program. The second study is a lab-based study that will take place in the Immersive Virtual Environment Testing Area in the NIH Clinical Center. In both studies, overweight, adult women will undergo a task designed to elicit mild-to-moderate emotional states. In Study 1 the elicited emotions will include anger, fear and neutral; Study 2 will include only anger and fear. Participants will then participate in a weight counseling encounter with a simulated doctor who will provide weight management information that includes discussions of either behavioral or genomic etiology. Participants in Study 1 will engage with the doctor via video clips over the internet, participants in Study 2 will engage with the doctor in an immersive virtual environment. Primary outcome measures pertain to participants health-related attitudes, behavioral intentions, and perceptions of stigmatization related to weight. Participants will include women who have a BMI of greater than or equal to 25. The final data set in Study 1 will include approximately 600 participants who are already part of an existing, nationally representative internet panel (ceiling n=700). The final data set in Study 2 will include approximately 250 participants recruited from the local area (ceiling n=500).

ELIGIBILITY:
* All participants will be adult women

INCLUSION CRITERIA ARE:

1. being between 18 and 50 years old;
2. having a self reported body mass index of greater than or equal to 25;
3. having the ability to read, write, and converse in English;
4. being able to come to the NIH Clinical Center for one visit.

EXCLUSION CRITERIA INCLUDE:

1. having a vestibular or seizure disorder;
2. having a high propensity for motion sickness;
3. known pregnancy;
4. uncorrected low vision or hearing;
5. inability to complete tasks in the virtual environment;
6. being or training to become a physician;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participants will be adult women. Inclusion for Study 1 are: (1) being part of a Knowledge Networks Panel; (2) having a self-reported body mass index of greater than or equal to 25. Inclusion criteria for Study 2 are: (1) being between 18 and 50 years old; (2) having a self-reported body mass index of greater than or equal to 25; (3) having the ability to read, write, and converse in English; (4) being able to come to the NIH Clinical Center for one visit.
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2013-07-05 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

PRIMARY OUTCOMES:
A | ongoing
  The primary goal of this research project is to continue building an evidence base on the benefits or pitfalls of introducing genomic information into weight-related primary care encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tetlock PE, Kristel OV, Elson SB, Green MC, Lerner JS. The psychology of the unthinkable: taboo trade-offs, forbidden base rates, and heretical counterfactuals. J Pers Soc Psychol. 2000 May;78(5):853-70. doi: 10.1037//0022-3514.78.5.853. PMID 10821194
- [Background] Agurs-Collins T, Khoury MJ, Simon-Morton D, Olster DH, Harris JR, Milner JA. Public health genomics: translating obesity genomics research into population health benefits. Obesity (Silver Spring). 2008 Dec;16 Suppl 3(Suppl 3):S85-94. doi: 10.1038/oby.2008.517. PMID 19037221
- [Background] Kushner RF. Understanding obesity by asking the right questions. Perspect Biol Med. 2010 Winter;53(1):148-51. doi: 10.1353/pbm.0.0139. PMID 20201162
- [Derived] Persky S, Ferrer RA, Klein WM. Nonverbal and paraverbal behavior in (simulated) medical visits related to genomics and weight: a role for emotion and race. J Behav Med. 2016 Oct;39(5):804-14. doi: 10.1007/s10865-016-9747-5. Epub 2016 May 4. PMID 27146511
- [Derived] Persky S, Ferrer RA, Klein WM. Genomic Information may Inhibit Weight-Related Behavior Change Inclinations Among Individuals in a Fear State. Ann Behav Med. 2016 Jun;50(3):452-9. doi: 10.1007/s12160-016-9771-2. PMID 26850762
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-HG-0158.html